CLINICAL TRIAL: NCT04259281
Title: A Phase 1/2 Open-label, Multiple-dose, Dose-escalating Clinical Trial of the Safety and Tolerability of GTX-102 in Pediatric Patients With Angelman Syndrome (AS)
Brief Title: A Study of the Safety and Tolerability of GTX-102 in Children With Angelman Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GTX-102-001; 2021-001793-36 (EudraCT Number)
Record Dates: First submitted 2020-01-31; First posted 2020-02-06 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Angelman Syndrome
MeSH Terms: conditions — Angelman Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- GTX-102 Cohort 1 (Experimental): 3.3 mg starting dose followed by intra-patient dose escalation up to 36 mg and then a maintenance phase (in U.S participants 4 to <17 years of age)
  Interventions: Drug: GTX-102
- GTX-102 Cohort 2 (Experimental): 10 mg starting dose followed by intra-patient dose escalation up to 36 mg and then a maintenance phase (in U.S participants 4 to <17 years of age)
  Interventions: Drug: GTX-102
- GTX-102 Cohort 3 (Experimental): 20 mg starting dose followed by intra-patient dose escalation up to 55 mg and then a maintenance phase (in U.S participants 4 to <17 years of age)
  Interventions: Drug: GTX-102
- GTX-102 Cohort 4 (Experimental): 3.3 mg starting dose followed by slow intra-patient dose escalation up to 5 mg and then a maintenance phase (in Ex-U.S participants 4 to <8 years of age)
  Interventions: Drug: GTX-102
- GTX-102 Cohort 5 (Experimental): 5 mg starting dose followed by slow intra-patient dose escalation up to 7.5 mg and then a maintenance phase (in Ex-U.S participants ≥ 8 to 17 years of age)
  Interventions: Drug: GTX-102
- GTX-102 Cohort 6 (Experimental): 7.5 mg starting dose followed by slow intra-patient dose escalation up to 10 mg and then a maintenance phase (in Ex-U.S participants 4 to <8 years of age)
  Interventions: Drug: GTX-102
- GTX-102 Cohort 7 (Experimental): 10 mg starting dose followed by slow intra-patient dose escalation up to 12 mg and then a maintenance phase (in Ex-U.S participants ≥ 8 to 17 years of age)
  Interventions: Drug: GTX-102
- GTX-102 Cohort US (Experimental): 2 mg for 4 monthly doses followed by a quarterly maintenance regimen
  Interventions: Drug: GTX-102
- GTX-102 Expanded Enrollment Cohort A (Experimental): Sponsor selected dose followed by slow intra-patient dose escalation and then a maintenance phase (in Ex-U.S participants 4 to <8 years of age)
  Interventions: Drug: GTX-102
- GTX-102 Expanded Enrollment Cohort B (Experimental): Sponsor selected dose followed by slow intra-patient dose escalation and then a maintenance phase (in Ex-U.S participants ≥ 8 to 17 years of age)
  Interventions: Drug: GTX-102
- GTX-102 Expanded Enrollment Cohort C (Experimental): Sponsor selected dose followed by slow intra-patient dose escalation and then a maintenance phase (in U.S participants 4 to <8 years of age)
  Interventions: Drug: GTX-102
- GTX-102 Expanded Enrollment Cohort D (Experimental): Sponsor selected dose followed by slow intra-patient dose escalation and then a maintenance phase (in U.S participants ≥ 8 to 17 years of age)
  Interventions: Drug: GTX-102
- GTX-102 Cohort E (Experimental): Sponsor selected dose followed by slow intra-patient dose escalation and then a maintenance phase (in participants that transition from GTX-102 US Cohort only)
  Interventions: Drug: GTX-102

INTERVENTIONS:
Drug: GTX-102 — antisense oligonucleotide

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of multiple-ascending doses of GTX-102 administered by intrathecal (IT) injection to participants with Angelman Syndrome (AS).

DETAILED DESCRIPTION:
This is a Phase 1/2, open-label, multiple-dose, study to evaluate the safety, tolerability, and plasma and CSF concentrations of GTX-102 in pediatric participants with AS.

The study includes a Loading phase followed by a Maintenance phase. Participants may continue on GTX-102 during the Maintenance phase of the study until GTX-102 is commercially available, intolerable toxicity occurs, the parent/legal guardian withdraws consent, the participant enrolls in another experimental study, or this study is terminated.

This study was previously posted by GeneTX Biotherapeutics, LLC and was transferred to Ultragenyx in July 2022.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from parent(s) or legal guardian(s)
* Documented genetic confirmation of full maternal UBE3A gene deletion causing AS in the region of 15q11.2-q13 including class I, II or III
* Stable seizure control (defined as clinically stable with no changes in antiepileptic medications over the prior 1 month before the screening visit, other than weight associated dose adjustments)
* Able to ambulate independently, or with an assistive device (note, a child whose primary means of mobility is by wheelchair is excluded from the study)
* Platelet count, prothrombin time / international normalized ratio, and partial thromboplastin time within 1.2 x the normal limits
* Normal renal function with serum creatinine and spot urine protein ≤ 1.4 x the upper limit of normal (ULN)
* Normal hepatic function with total bilirubin, aspartate aminotransferase, alanine aminotransferase, and alkaline phosphatase ≤ 1.4 x ULN. Exception: levels ≤ 2 × ULN are acceptable if due to anti-epileptic drugs (AEDs) or Gilbert syndrome
* Willing and able to comply with scheduled visits, drug administration plan, laboratory tests, study restrictions, and all study procedures, including LP procedure
* Able to tolerate the anesthetic regimen, if required for LP procedure
* A female patient is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: Female of non-childbearing potential (ie, pre-menarche), Female of childbearing potential who agrees to remain abstinent (refrain from heterosexual intercourse) or use acceptable contraceptive methods during the treatment period and for at least 3 months after the final dose of GTX-102
* A male patient is eligible to participate if he agrees to remain abstinent (refrain from heterosexual intercourse) or use acceptable contraceptive methods during the treatment period and for at least 3 months after the final dose of GTX-102

Exclusion Criteria:

* Any change in medications (excluding AEDs) or diet/supplements intended to treat symptoms of AS (eg, sleeping aids, supplements, dietary change including ketogenic or low-glycemic index diet, other) over the prior 1 month before screening
* Any bleeding or platelet disorder
* Any clinically significant cardiovascular, endocrine, hepatic, renal, pulmonary, gastrointestinal, neurological, malignant, metabolic, psychiatric, or other condition that, in the judgment of the Investigator, will pose a safety risk, make the patient unsuitable for participation in, and/or unable to complete the study procedures
* Any laboratory abnormality, that, in the Investigator's opinion, could adversely affect the safety of the patient, make it unlikely that the course of treatment or follow up would be completed, or impair the assessment of study result
* Known positive for hepatitis B virus, hepatitis C virus, or human immunodeficiency virus
* Any active infection
* Bone, spine, bleeding, or other disorder that exposes the patient to risk of injury or unsuccessful lumbar puncture
* Drugs that increase the risk of bleeding (eg, heparin, low molecular weight heparin, platelet inhibitors)
* Any prior use of gene therapy
* Use of any investigational drugs in the past 6 months or within 5 half-lives, whichever period is greater (with the exception of prior GTX 102)
* Known hypersensitivity to any oligonucleotide, as demonstrated by an immune mediated reaction (eg, pneumonitis, hepatitis, nephritis, neuritis, or other system inflammation), or a systemic allergic reaction such as signs and symptoms of anaphylaxis, urticaria, clinically significant rash
* Patient is pregnant or lactating
* Any medical condition that would require intubation for the anesthesia procedure

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs), Serious AEs (SAEs), Adverse Events of Special Interest (AESIs), AEs Leading to Discontinuation and Severity of AEs | Up to Day 337

SECONDARY OUTCOMES:
Pharmacokinetics of GTX-102 over time | Up to Day 337
  Maximum drug concentration (Cmax)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (25):
- United States (6):
  - UCLA Medical Center, Los Angeles, California
  - Rady Children's Hospital, San Diego, California
  - Rare Disease Research, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Weill Cornell Medicine, New York, New York
- Australia (3):
  - Austin Health, Heidelberg, Victoria
  - The Royal Children's Hospital, Parkville, Victoria
  - Queensland Children's Hospital, South Brisbane
- Canada (5):
  - MAGIC Clinic Ltd, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - McGill University Health Centre, Montreal, Quebec
- France (2):
  - Hopital de la Timone, Marseille
  - AP-HP Hopital Necker-Enfants Malades, Paris
- Germany (2):
  - Universitatsklinikum Leipzig, Leipzig, Saxony
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
- The Edmond and Lily Safra Children's Hospital, Ramat Gan, Israel
- Spain (3):
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Barcelona
  - Hospital Universitari Parc Tauli, Sabadell, Barcelona
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
- United Kingdom (3):
  - Cambridge University Hospitals, Cambridge
  - Great Ormond Street Hospital for Children, London
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dindot SV, Christian S, Murphy WJ, Berent A, Panagoulias J, Schlafer A, Ballard J, Radeva K, Robinson R, Myers L, Jepp T, Shaheen H, Hillman P, Konganti K, Hillhouse A, Bredemeyer KR, Black L, Douville J; FIRE consortium; FIRE Consortium. An ASO therapy for Angelman syndrome that targets an evolutionarily conserved region at the start of the UBE3A-AS transcript. Sci Transl Med. 2023 Mar 22;15(688):eabf4077. doi: 10.1126/scitranslmed.abf4077. Epub 2023 Mar 22. PMID 36947593